CLINICAL TRIAL: NCT06932406
Title: Orofacial Pain Self-management: Personality Moderation Effect - Randomized Clinical Trial
Brief Title: Orofacial Pain Self-management: Personality Moderation Effect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCV/2023-2024/072
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-01

CONDITIONS: Chronic Orofacial Pain; Temporomandibular Disorder (TMD); Temporomandibular Disorders (TMD); Temporomandibular Dysfunction (TMD)
Keywords: Temporomandibular disorder; Orofacial pain; Self-management; self-efficacy; therapeutic exercise; therapeutic education; cognitive behavioral; mind-body techniques; Lifestyle modification training; manual therapy; personality; psychosocial; biopsychosocial; physiotherapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Intervention Model Description: A prospective, longitudinal, comparative randomized clinical trial (RCT) will be conducted. The sample will be composed of adults with chronic orofacial pain who meet the inclusion and exclusion criteria of the study. Three measurements will be performed: pre-intervention, post-5 weeks and post-6 months. The study is based on the principles of the 2017 Declaration of Helsinki, all participants will be informed at all times and prior to study participation will be required to sign informed consent. The intervention design has been designed based on the CONSORT Guidelines for Randomised Clinical Trials and will be registered on ClinicalTrials.gov.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management Group (Experimental): This group will implement a protocol based on self-management consisting of 5 levels of strategy: educational concepts and dynamics, cognitive behavioural tools, therapeutic exercise of the orofacial region, guidelines and strategies for lifestyle modification and mindbody tools. This protocol was developed by conducting a previous Scoping Review abouts application methods of selfmanagement in orofacial region. The intervention will be carried out in 5 total sessions of 45-60 minutos over 10 weeks.
  Interventions: Other: Self-management intervention
- Clinical Practice Guideline Group (Active Comparator): The protocol will be based on the Clinical Practice Guideline for the Management of Temporomandibular Disorders 2021. Following the guideline, there will be 5 sessions of pathology and pain education, cognitive behavioural tools for bruxism and parafunctional habits, jaw exercises for motor control, mobility and strength, and manual therapy. The intervention will be carried out in 5 total sessions of 45-60 minutos over 10 weeks.
  Interventions: Other: Clinical Practice Guideline Intervention

INTERVENTIONS:
Other: Self-management intervention — This intervention will implement a self-management protocol. It will consist in 5 strategy levels: educational concepts and dynamics, cognitive behavioural tools and processes, therapeutic exercise of the orofacial region, guidelines and strategies for lifestyle modification and mindbody tools.
  Several of the above 5 strategies will be employed in each session. Education will include TMD concepts, pain neurophysiology, contextualisation of pain in terms of perceived stress, anxiety and others. Exercises will aim to train motor control, strength and mobility. Cognitive behavioural tools will be used to modulate pain relationship through behaviour modification. Processes such as cognitive distraction, gradual exposure to movement or the scheduling of self-care activities will be used. Mindbody strategies such as relaxation exercises and pain acceptance will seek to reduce the patient's frustration with pain. Structured guidelines will be included to achieve desirable lifestyle changes.
  Other Names: GSelf-Management; GS-M
  Arms: Self-management Group
Other: Clinical Practice Guideline Intervention — Following the guidelines, 5 sessions of education, cognitive behavioural tools, jaw exercises and manual therapy will be conducted.
  The educational sessions will teach about TMD and basic pain concepts. A single type of cognitive behavioural tool will be employed. The aim will be to decrease bruxing and parafunctional activity during wakefulness. This will be done by training the jaw relaxation position, which will then be generalised to activities of daily living with the help of some conditioning through positive and negative reinforcement. Exercise activities will aim to train motor control, strength and mobility. Manual therapy will be carried out in the orofacial region by means of soft tissue techniques and joint mobilisation.
  Other Names: GClinical Practice Guideline; GCPG
  Arms: Clinical Practice Guideline Group

SUMMARY:
The objective of this clinical trial is to study the effect of self-management on pain perception in patients with chronic orofacial pain and temporomandibular disorders (TMD) comparing it with the conventional treatment proposed by the TMD clinical practice guidelines. It also evaluates its effect on function and various psychosocial variables.

As a secondary objective, this work proposes to study the variability between patients, in terms of personality factors, as moderators of the effect of treatment on pain perception. Including in the proposed statistical models certain covariates such as perception and/or coping with stress, anxiety and other psychosocial variables.

This is a randomized clinical trial with two intervention groups and three measurement times (T0; pre-intervention, T1; post-5 weeks and T2; post-6 months). The experimental group will be applied a protocol based on self-management, which includes: therapeutic education, cognitive-behavioral tools, therapeutic exercise of the temporomandibular region, mind-body strategies and modifications of aspects related to lifestyle. The control group will carry out an intervention program based on the Clinical Practice Guidelines for the Management of Temporomandibular Joint Disorders. Therefore, using a set of tools based on therapeutic education, cognitive-behavioral tools for bruxism and other parafunctional habits, temporomandibular region exercises and manual therapy.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are the most common cause of chronic orofacial pain and encompass a range of syndromes affecting the masticatory muscles and temporomandibular joints (TMJ). Approximately 9-13% of the population experiences orofacial pain related to TMD. The high complexity, multifactorial nature, recurrence, and long duration of chronic pain increase the need for approaches focused on a multi-component management, based on learning strategies and coping skills, self-efficacy, and self-care. These approaches can be classified as self-management interventions, and their multifactorial nature makes them suitable for application and teaching by various health professionals. Within this multifactoriality, previous studies have shown that the patient's personality influences the occurrence and progression of chronic pain. The objective of this study is to evaluate a comprehensive self-management program in patients with chronic orofacial pain to assess its effect on pain perception and other psychosocial and functional variables, and subsequently analyze the moderation of factors related to the patient's personality on the intervention outcomes.

It is hypothesized that the self-management-based treatment is effective in reducing pain perception in the short and medium term, and that personality is a moderating factor for the intervention's effect.

The study will be conducted on 98 subjects aged 18 to 65, diagnosed with TMD and chronic orofacial pain. The intervention will last for 10 weeks with 5 sessions of application and 3 sessions of evaluation (pre-intervention; during the session time for the first intervention application session, post-5 weeks during the session time for the last intervention application session, and post-6 months; in an extra session dedicated solely to making the evaluation record). Each intervention session will be held once every two weeks. Results will be assessed using the EVA and GCPS questionnaires (pain), PCS (catastrophizing), TSK/TMD/S (kinesiophobia), FABQ (fear-avoidance), MFIQ (mandibular dysfunction), CPSS (self-efficacy), MMO (mandibular opening), Borg (perceived fatigue), BFQ (personality), CLCD (pain locus), COPE28 (stress coping), PSS (stress perception), STAI (anxiety), pressure algometry (pain threshold), intra-articular sound quantification, and treatment-seeking behavior.

All variables will be taken in triplicate at all three measurement times with the exception of the personality-related variable (BFQ). A descriptive statistical analysis of all variables in each of the intervention groups will be performed. To analyse the effect of the intervention on pain and the other secondary variables, a repeated-means ANOVA analysis will be performed between the self-management group (GSelfManagement) and the group based on the clinical practice guideline (GGuide). To examine whether variation in pain at follow-up is influenced by personality variables and/or the psychosocial variables kinesiophobia, catastrophising thoughts, fear-avoidance, type of pain control, perception of stress and anxiety, and stress coping, a moderation and mediation analysis will be performed. This analysis determines whether the effect size of a causal variable X (VAS and GCPS, MFIQ, MMO and VAS Fatigue) on outcome Y (GGuide and GSelfManagement), depends on a moderating or mediating variable W (i.e., kinesiophobia, catastrophizing, fear-avoidance, stress and anxiety perception, stress coping, personality and type of pain control). The degree of significance will be set at p<0.05. All analyses will be performed using statistical analysis software (SPSS 24 Inc, Chicago, Illinois, USA and The PROCESS macro for SPSS).

ELIGIBILITY:
Inclusion Criteria:

* The patient presents TMDs diagnosed according to the CD/TMD classification.
* Age between 18 and 65.
* Presence of pain in mandibular, temporal, facial, peri-auricular and/or auricular regions.
* Presence of chronic orofacial pain. Defined by the ICD-11 as orofacial pain or headache that occurs for more than two hours a day for 50% of the days of the last three months.
* Orofacial pain is related to TMDs according to the International Classification of Headaches.
* Moderate pain intensity, corresponding to a weekly average of at least 30 mm on a 100 mm VAS (validated representation of moderate pain on the VAS scale = 31-54 mm)

Exclusion Criteria:

* Concomitant rheumatic systemic pathologies.
* History of trauma or recent surgical intervention in the head, face, neck or chest.
* Presence of intraoral infections or odontogenic pain.
* Headache of neuropathic origin (trigeminal neuralgia, Arnold neuralgia, etc.).
* Being receiving therapy (except rescue pharmacological therapy) for this disorder or pain.
* Cognitive impairment that prevents the follow-up of an educational program (determined through the MoCA questionnaire)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-05-24 (Estimated); Study Completion 2026-05-24 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  Pain intensity assessment instrument consisting of a 10-centimetre horizontal line numbered from 0 to 10, where 0 represents no pain and 10 represents the greatest unimaginable pain. The patient must mark on the line the point that indicates the intensity of his or her pain and then it is measured with a millimetre ruler. The intensity is expressed in centimetres or millimetres. If reporting a score on this scale, it is important to include the minimum and maximum values (0 and 10, respectively), as well as clarify that higher scores represent worse pain intensity. This tool has a high reliability, with an Internal Consistency (IC) of 0.97.
Chronic Pain Grading Scale 2.0 Spanish Version (GCPS) | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  Quantitative assessment scale of chronic pain that evaluates the degree of pain using 8 items, quantifying the number of days of pain in the last 6 months, current pain, average and maximum monthly pain and pain and limitation in ADL, social and occupational activities. Each item measures the score on an 11-point Likert scale, with a total range from 0 to 70 points. The tool has an internal consistency, represented by Cronbach's α coefficient, of 0.87 (95% CI, 0.83-0.92). If reporting a score on this scale, it is important to include the minimum and maximum values (0 and 70, respectively), as well as clarify that higher scores represent worse outcomes.

SECONDARY OUTCOMES:
Demographic data | These data will be collected pre-intervention.
  A standardised questionnaire will be used to collect information on age, sex, profession, concomitant conditions, drugs used (number, name and category).
Pain Catastrophizing Scale (PCS) | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  A scale that assesses catastrophic thoughts, consisting of 3 dimensions: rumination (constant worry and inability to inhibit pain-related thoughts), magnification (exaggeration of the unpleasantness of pain situations and expectations of negative consequences) and helplessness (inability to cope with painful situations). It consists of 13 items with a five-point Likert-type response scale (0 = Not at all; 4 = All the time), with scores ranging from 0 to 52. High scores indicate a greater presence of catastrophic thoughts.
  This tool has an internal consistency (Cronbach's α) of 61.8%->70%.
The Tampa Scale of Kinesiophobia for Temporomandibular Disorders Versión Español (TSK11-TMD-S) | It will be used in pre-intervention, post-5 weeks and post-6 months analyses.
  Scale assessing kinesiophobia or fear of movement or injury in patients with TMD.
  The scale consists of a total of 11 items. In each of the items, the user must indicate his or her degree of agreement with each of the statements presented. In this way, it is scored using a Likert-type scale from 1 (totally disagree) to 4 (totally agree), with higher scores being indicators of greater fear of movement.
  It has an Internal Consistency (Cronbach's α) of 0.843.
Fear-Avoidance Beliefs Questionnaire (FABQ) | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  It is a self-administered questionnaire that assesses the patient's fear-avoidance beliefs about physical activity and work. It assesses activities of daily living, behaviour, functional mobility, general health, participation, mental health, motivation, occupational performance, pain, personality, quality of life, self-efficacy, stress and coping. It consists of 16 items in which the patient scores his or her degree of agreement or disagreement with the statement proposed in each item, using a 7-point Linkert-type scale. Where 0 symbolises complete disagreement and 6 complete agreement. The maximum score that can be obtained is 96 points, with higher scores indicating higher fear-avoidance beliefs. It consists of two subscales: the work subscale (FABQw) with 7 questions and a maximum score of 42 points, and the physical activity subscale (FABQpa) with 4 questions and a maximum score of 24.
  ICC=0.97,FABQpa CI=0.77,FABQw=0.88. The total maximum score that can be obtained is 96 points
The Mandibular Function Impairment Questionnaire (MFIQ) | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  To assess the perception of jaw function. Consists of two dimensions of 17 items in total that assess the degree of disability of various specific jaw functions. Each item is scored on a scale from 0 to 4, where 0 represents no difficulty and 4 represents extreme difficulty in performing a specific task. The sum results in a scale from 0 to 68, where higher scores represent a greater degree of disability.
  The overall Internal Consistency of the scale is Cronbach's α =0.94, with Cronbach's α =0.87 for the first dimension and Cronbach's α =0.92 for the second dimension.
Máxima apertura de la boca (MMO) | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  Quantification of the maximum jaw opening distance by measuring the upper and lower interincisive space during maximum jaw opening with a caliper (in millimetres). Three consecutive measurements shall be taken and the average of the three shall be recorded. It shall be measured in two ways: active maximum mandibular opening (MMO) and comfortable maximum opening (MCO). This type of measurement is frequently used in other similar articles.
Intra-articular sounds | To be used in pre-intervention, post-5 weeks and post-6 months analyses.
  The presence and type of intra-articular sounds will be confirmed pre-intervention by the investigator collecting the data using a stethoscope placed over the mandibular condyle during the exploration of TMJ movement.
  The procedure used to subjectively analyse intra-articular sounds has been described in other studies previously. To quantify the intensity of intra-articular sounds a numerical scale (NRS 0-10) will be used, the frequency will be reported by selecting one of the following options: 0 No joint sounds, 1 Joint sounds once or twice/week, 2 Joint sounds three/four times per week, 3 Joint sounds ≥ five times/week.
Borg Scale | It will be collected during each of the exercise sessions to check compliance with the intensity of the exercises. The data will not be processed statistically.
  Exercise fatigue will be assessed using the Borg Scale, which has been used in other research to measure fatigue in different physical exercise contexts. This scale of perceived exertion measures the degree of effort that the individual perceives when doing a given exercise on a numerical scale from 0 to 10, where 0 is total rest and 10 is maximum effort. This tool will be used during each of the exercise sessions to ensure that the programmed intensity is met.
Big Five Personality Test (BFQ) | This tool will be used in the pre-intervention measurement.
  The Big Five (BFQ) is a five-factor model to describe personality.. It uses a Likert-type scale consisting of 132 questions with five response options ranging from 'completely false for me' to 'completely true for me'. It identifies the five fundamental dimensions for describing and assessing personality (open-mindedness, emotional stability, responsibility, agreeableness, energy) and their respective sub-dimensions (openness to experience, openness to culture, impulse control, emotion control, perseverance, conscientiousness, friendliness, cooperation, dominance, dynamism). The Internal Consistency of Cronbach's alpha test has a significant value of 0.874 for the five scales and the ten subscales. When reporting a score on the BFQ, the total score ranges from 132 to 660, with higher scores indicating greater alignment with the positive characteristics of each personality dimension. Higher scores generally reflect better outcomes in terms of personality traits associated with positive
Pain Locus of Control Questionnaire (CLCD) | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  The instrument consists of 33 items divided into three subscales assessing: (a) internal locus of control, which refers to people's beliefs about whether their pain is influenced by personal actions ('I can prevent pain if I avoid certain situations that make me nervous'; Cronbach's α = 0. 86); (b) locus of control by chance, determined by the degree to which a person believes that their pain is due to chance ('my pain cannot be controlled'; Cronbach's α = 0.84); and (c) locus of control by health professionals under the belief that their pain will be relieved by health professionals ('my doctor's treatment can help me reduce my pain'; Cronbach's α = 0.88). Responses to the instrument were made on a five-point scale, ranging from strongly disagree to strongly agree. Higher scores on the scale indicate a stronger belief in control over pain through internal factors, health professionals, or chance, depending on the subscale.
Pressure Algometry | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses
  The pressure algometer is an instrument with a circular disc on which the pressure measurements are displayed (with a range of 5 kg, divided into 10 parts of half a kilogram), and a rubber tip with a circular surface of 1 cm2, which allows the pressure force to be transferred to deep tissues. The FPK 60 Analogue Algometer will be used in this study.
  Its application follows the protocol proposed by another similar study. The tip of the algometer will be applied perpendicular to the muscle and a pressure will be maintained, progressively increasing at 1 kg/sec. Subjects will be instructed to make a signal at the moment they experience pain, in order to have an accurate record (pain threshold). The points where algometry will be performed are: masseter, temporalis and trapezius muscles and the suboccipital level.
The SCL-90-R Symptom Inventory | It will be used in the pre-intervention analysis.
  This inventory was developed to assess patterns of psychosocial symptoms present in individuals, and can be used in both community tasks and clinical diagnosis. Each of the 90 items is answered on a five-point scale (0-4). It is assessed and interpreted according to nine primary dimensions and three global indices of psychological distress: (1) somatizations (SOM), (2) obsessions and compulsions (OBS), (3) interpersonal sensitivity (SI), (4) depression (DEP), (5) anxiety (ANS), (6) hostility (HOS), (7) phobic anxiety (FOB), (8) paranoid ideation (PAR), (9) psychoticism (PSIC) and other indices such as (1) global severity index (GSI), (2) total positive symptoms (TSP) and (3) positive symptomatic distress index (PSDI). In spanish population; CI=0.72-0-96, in terms of chronic pain; CI=0.78-0,97. Higher scores on this inventory indicate more significant psychosocial symptoms and distress, which may be relevant in diagnosing psychological conditions or assessing the impact of chronic pain
Brief Coping Coping with Stress Questionnaire (COPE28) | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  A multidimensional inventory, developed to assess different forms of stress coping. Five of its scales (four items each) conceptually measure different aspects of problem-focused coping (active coping, planning, suppression of distracting activities, restraining coping, seeking instrumental social support). This scale has an Internal Consistency of between 0.71 and 0.80 as measured by Cronbach's alpha. Minimum score: 0 (indicating no use of the particular coping strategy). Maximum score: 4 (indicating maximum use of the coping strategy).
The Perceived Stress Scale (PSS) questionnaire. | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  A self-report instrument that assesses the level of perceived stress over the past month, it consists of 14 items with a five-point scale response format (0 = never, 1 = hardly ever, 2 = occasionally, 3 = often, 4 = very often). The total PSS score is obtained by inverting the scores of items 4, 5, 6, 7, 9, 10 and 13 (as follows: 0=4, 1=3, 2=2, 3=1 and 4=0) and then adding the 14 items. The direct score obtained indicates that a higher score corresponds to a higher level of perceived stress. This scale has an Internal Consistency of 0.81 and a test-retest validity of 0.73. Higher scores indicate a higher level of perceived stress in the past month. Lower scores suggest that the individual has experienced lower levels of perceived stress.
The Strait Anxiety Questionnaire (STAI) | It will be used in the pre-intervention, post-5 weeks and post-6 months analyses.
  A questionnaire intended to assess individuals' anxiety level. More specifically, the STAI measures individuals' predisposition to perceive various stimuli as threatening (i.e. trait anxiety). Thus, an individual with high trait anxiety is more likely to produce an anxiety response. It includes 40 items (i.e. 20 for each subscale), the response scale ranges from 0 to 3 points. In the State Anxiety subscale, item scores range from 0=not at all [not at all], 1=somewhat [somewhat], 2=quite a bit [moderately], and 3=very much [a lot]. In the Trait Anxiety subscale, response options range from 0=almost never [almost never], 1=sometimes [sometimes], 2=often [often], and 3=almost always [almost always]. Although each subscale has a theoretical range of 20 to 80, the scores can be compared with those of the original scale by adding 20 to the scores obtained.The Cronbach's alpha for this scale is 0.82. Higher scores on either subscale indicate higher levels of anxiety.

OTHER OUTCOMES:
Treatment adherence | This variable will be collected post 5 weeks and reviewed during the treatment.this variable will not be used in this disc analysis
  Defined by the WHO as 'the degree to which a patient's behaviour, in relation to taking medication, following a diet or modifying lifestyle habits, corresponds to the recommendations agreed with the health professional'.
  Participants will be given a diary-like notebook to fill in with the activities carried out on a weekly basis. This method of recording adherence to therapeutic exercise has been used previously in other studies. Each patient will be warned that failure to complete a minimum number of activities (70%) will result in exclusion from the study.
Montreal Cognitive Assessment Test (MoCA Test) | This variable will be collected pre-intervention as a measure to objectify the absence of cognitive impairment and to justify the part related to cognitive abilities that allow the patient to be included in the study. It will not be treated for statistic
  A brief screening test for the identification of mild cognitive impairment and early dementia processes. The total score of the MoCA test is 30 points, and the administration time is 7-10 ms. It is validated in the Spanish population between 18 and 90 years of age. It assesses the general cognitive status of the individual through different cognitive domains. Total score: The maximum score is 30 points, and the minimum score is 0 points. A higher score indicates better cognitive functioning, while a lower score suggests a higher likelihood of cognitive impairment. Typically, a score below 26 points may indicate possible cognitive impairment, though interpretation should consider other factors such as education level and clinical context.
Self-reporting of educational level | This variable will be collected at the pre intervention time.
  The educational level was obtained through the question 'What is the highest level of education you have completed?', where 8 options could be selected (1. primary education or lower, 2. secondary education, 3. baccalaureate, 4. vocational training, 5. degree studies).

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Univerity of Valencia, Valencia, Valencia, Spain